CLINICAL TRIAL: NCT02433353
Title: Results From a 24 Week, Double-blind, Placebo-controlled Trial of EMDR Combined With Venlafaxine XR in the Treatment of Posttraumatic Stress Disorder
Brief Title: Results From a 24 Week Trial of EMDR Combined With Venlafaxine XR
Acronym: EMDRVEN
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: PI was transferred to another base. No one else available to serve as PI.
Sponsor: Bayne-Jones Army Community Hospital (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Bayne-Jones
Record Dates: First submitted 2015-04-09; First posted 2015-05-05 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Posttraumatic Stress Disorder
Keywords: PTSD; posttraumatic stress disorder; venlafaxine; EMDR; eye movement desensitization reprocessing; antidepressant; psychotherapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Venlafaxine Hydrochloride; Eye Movement Desensitization Reprocessing; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- EMDR + Venlafaxine XR (Experimental): Participants will receive 12 one-hour sessions of EMDR while taking venlafaxine XR 150mg or 225mg for the duration of the 6 month study.
  Interventions: Drug: Venlafaxine XR; Behavioral: EMDR
- EMDR + Placebo (Placebo Comparator): Participants will receive 12 one-hour sessions of EMDR while taking placebo 150mg or 225mg for the duration of the 6 month study.
  Interventions: Behavioral: EMDR; Drug: Placebo

INTERVENTIONS:
Drug: Venlafaxine XR — Serotonin norepinephrine reuptake inhibitor
  Other Names: Effexor
  Arms: EMDR + Venlafaxine XR
Behavioral: EMDR — psychotherapy
  Other Names: Eye Movement Desensitization Reprocessing
Drug: Placebo — Look-alike venlafaxine XR tablets containing no active drug
  Other Names: Sugar pill
  Arms: EMDR + Placebo

SUMMARY:
Approximately 150 active duty service members meeting Diagnostic and Statistical Manual version 5 (DSM-5) criteria for posttraumatic stress disorder (PTSD) and scoring 50 or above on the Clinician Administered PTSD Score for DSM-5 (CAPS-5) will be recruited. Qualifying participants will be randomized on a 1:1 basis to either the eye movement desensitization reprocessing (EMDR) plus venlafaxine XR group or the EMDR plus placebo group. Protocol will call for participants to complete 12 one-hour EMDR session while taking a venlafaxine XR/placebo dose of 150mg or 225mg for the entire 24 weeks. Both prescribers and therapists will be blinded and CAPS-5 assessments will be completed by an individual not involved in a participant's direct treatment. An unblinded pharmacist will dispense medication or placebo according the instructions of the prescriber and will count remaining tablets to measure compliance. All EMDR sessions will be recorded and will be reviewed by the principal investigator using a fidelity checklist. CAPS-5 will be administered after completion of EMDR and again at 6 months from the date of his/her first therapy session.

DETAILED DESCRIPTION:
Approximately 150 active duty service members meeting DSM-5 criteria for PTSD and scoring 50 or above on the Clinician Administered PTSD Score for DSM-5 (CAPS-5) will be recruited for a prospective, randomized, double-blinded, controlled trial. Participants will be recruited via referral from other providers or self-referral from recruitment fliers. CAPS-5 is considered the gold-standard for PTSD symptom assessment in research. An initial PHQ-9,PCL-5, urine drug screen, and pregnancy test will be obtained at that visit as well. Qualifying participants will then meet with a prescriber, review informed consent, draw a number for randomization, and complete the SCID-5. The participant will then meet with the pharmacist who will dispense either venlafaxine XR or placebo. Randomization will have occurred before any participants have been recruited. Randomization will consist of use of a random number generator to generate 150 numbers. The pharmacist will secretly assign half of the numbers to treatment and half to control. Numbers generated will be written on slips of paper and placed in opaque envelopes then placed in a box. Participants will then draw their own numbers and inform the researchers of the number drawn. The titration schedule for the venlafaxine XR/placebo will be 3 days at 37.5mg, 7 days at 75mg, then increasing to 150mg. The participant will meet with the prescriber after 4 weeks at 150mg to determine if an increase to 225mg is warranted based on the participants DSM-5 PTSD symptoms. Meetings with a prescriber will then occur monthly throughout the study unless side effects or other concerns require more frequent follow up. Prescriber visits will be scheduled for 30 minutes, however, visits could be completed in as little as five minutes if the medication is working well with no side effects, blood pressure remains at baseline, the participant remains adherent to both medication and therapy, and the participant raises no concerns. Participants will meet with the pharmacist on a monthly basis for pill counts. EMDR sessions will occur weekly if possible and not any less than once every 2 weeks. Two sessions are allowed in 1 week if the participant anticipates going to the field or otherwise being unavailable for regular visits. All EMDR sessions will be recorded using a camcorder and the principal investigator will review 10% of all therapy sessions (a minimum of 1 session per participant) using a fidelity checklist. CAPS-5 assessments will be completed by an individual not involved in a participant's direct treatment and will be administered after completion of EMDR and again at 6 months from the date of his/her first therapy session. A urine drug screen will be ordered with each CAPS-5. Missing data/participant drop out will be handled using last object carried forward. Comparisons between interventions will be computed using a student's T-test for single comparisons between groups or ANOVA when multiple comparisons/time points are involved. If at any point a participant requests a record of treatment, a summary of care will be provided.

ELIGIBILITY:
Inclusion:

* Initial CAPS-5 score of 50 or greater
* Meeting criteria for PTSD using DSM-5 criteria
* Open to active duty US service members of all genders, races / ethnicities, religions, sexual orientations, and marital statuses
* Participants can have a history of mild TBI, past or current substance abuse, nicotine dependence, chronic pain, migraines/headaches, and most other medical illnesses not specified in exclusion section
* Participants can be taking opiates, a sleep aid, and/or prazosin for an indication of PTSD nightmares provided dosing does not exceed 15mg (men) / 9mg (women). Dosing more than once per day is not permitted

Exclusion:

* Current suicidal or homicidal ideation
* Pregnancy
* Profound hearing loss
* HIV and AIDS
* Current chemotherapy
* Primary thought disorders
* Bipolar disorder or cyclothymia
* Current substance dependence (not including nicotine)
* Current use of bupropion above 150mg daily
* Current use of mirtazapine above 15mg daily
* Current use of an SSRI
* Current use of another SNRI
* Current use of tricyclic antidepressants in doses above 50mg
* Current use of an MAO-I
* Current use of a stimulant
* Current use of a mood stabilizer/anti-epileptic for an indication of mood stability or reduction in anger
* Current use of an anti-psychotic
* Current use of lithium
* Chronic daily use of steroids
* Current use of tapentadol
* Current use of dronabinol
* Current use of ketamine

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change in PTSD symptoms at 12 weeks measured using the CAPS-5 scale | 12 weeks
  Clinician Administered PTSD Scale for DSM-5
Change in PTSD symptoms at 24 weeks measured using the CAPS-5 scale | 24 weeks
  Clinician Administered PTSD Scale for DSM-5

SECONDARY OUTCOMES:
Change in depression symptoms at 12 weeks measured using the PHQ-9 scale | 12 weeks
  Periodic Health Questionnaire
Change in depression symptoms at 24 weeks measured using the PHQ-9 scale | 24 weeks
  Periodic Health Questionnaire
Percentage of participants experiencing adverse events as a measure of safety and tolerability | 24 weeks
Attrition percentage as a measure of safety and tolerability | 24 weeks
Change in PTSD symptoms at 12 weeks measured using the PCL-5 scale | 12 weeks
  PTSD Checklist for DSM-5
Change in PTSD symptoms at 24 weeks measured using the PCL-5 scale | 24 weeks
  PTSD Checklist for DSM-5
Presence of non-prescribed or illicit drugs on urine drug screen at 12 weeks | 12 weeks
Presence of non-prescribed or illicit drugs on urine drug screen at 24 weeks | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Lee, MD, Principal Investigator — Bayne-Jones Army Community Hospital